CLINICAL TRIAL: NCT05503641
Title: Cognitive and Psychomotor Stimulation in the Physical and Cognitive Function and in the Functional Capacity of Older Adults
Brief Title: Cognitive and Psychomotor Stimulation in the Physical and Cognitive Function in the Functional Capacity of Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: - University of Jaén
Record Dates: First submitted 2022-08-13; First posted 2022-08-17 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This group receives training in cognitive and psychomotricity stimulation activities.
  Interventions: Other: Cognitive and psychomotor stimulation
- Control group (No Intervention): This group does not receive any treatment.

INTERVENTIONS:
Other: Cognitive and psychomotor stimulation — Each cognitive stimulation session aimed to maintain and/or improve cognition through memory, language, executive functions, attention, concentration, and perception activities. All the people in the two groups performed the same cognitive stimulation activities adapted to their cognitive and sensory abilities.
  The psychomotricity sessions were aimed at maintaining and/or improving the motor, cognitive, social and affective functioning of the person through activities that work on postural tone, body scheme, laterality, fine and gross motor skills, balance, flexibility, among others, adding a cognitive component. All the psychomotricity activities were adapted to the motor and cognitive abilities of the users.
  Arms: Experimental group

SUMMARY:
The population is increasingly older and this means that there are more and more dependent older people, for this reason it is necessary to achieve the best quality of life for the older adult population by promoting active and healthy aging.

ELIGIBILITY:
Inclusion Criteria:

* Have a mild dependency according to the Barthel Index (score greater than 60 points).
* Not present serious cognitive impairment, nor serious psychiatric or somatic disorders, nor disruptive and inappropriate behaviors.
* Be able to understand each of the self-administered questionnaires and perform the tests.

Exclusion Criteria:

* Have vision problems.
* Be enrolled in a physical exercise program.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Tinetti Scale | Up to twelve weeks
  Scale for the assessment of gait and balance. Indicated for early detection of the risk of falls in the elderly. The higher the score, the lower the risk of falls. The maximum score for the gait subscale is 12, for the balance subscale 16. The sum of both scores for the risk of falls.
Handgrip Strength | Up to twelve weeks
  Dynamometer will be employed to assess handgrip strength.
MMSE (mini-mental state examination) | Up to twelve weeks
  A tool that can be used to systematically and thoroughly assess mental status.
TUG test (Timed Up and Go test) | Up to twelve weeks
  Is a simple test used to assess a person's mobility and physical function.
The Lawton & Brody scale | Up to twelve weeks
  Evaluates independence and functionality in instrumental activities of daily life) such as shopping, cooking, cleaning, washing, finances, medication, transportation and use of the telephone; and considers instrumental disability the inability to perform one or more activities. Each area is scored according to the description that best corresponds to the subject. Therefore, each area scores a maximum of 1 point and a minimum of 0 points. The maximum dependence would be marked by obtaining 0 points, while a sum of 8 points would express total independence.
The Barthel Index | Up to twelve weeks
  Assesses functional dependence when performing basic activities of daily living (BADL), consists of 10 items with scores between 0 and 15 maximum each (Mahoney and Barthel, 1965). The highest possible score is 100 points, this being the greatest independence, if the score is greater than 60 the dependency is slight, if the score is between 40 and 55 the dependency is moderate, when between 20 and 35 points the dependency is serious and if it is less than 20 points the dependency is total.

SECONDARY OUTCOMES:
BMI (Body Mass Index) | Up to twelve weeks
  Is calculated from the formula, Weight (kg) / Height2 (m2), whose unit is kg/m2. It is a rough indicator of total body fat.
Body Weight | Up to twelve weeks
  Is the sum of Body Fat and Fat Free Mass.
Height | Up to twelve weeks
  It measures a person's height, measured from the sole of the foot to the top of the head.

CONTACTS AND LOCATIONS:
Locations (1):
- U.E.D. Virgen de la Capilla, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castellote-Caballero Y, Carcelen Fraile MDC, Aibar-Almazan A, Afanador-Restrepo DF, Gonzalez-Martin AM. Effect of combined physical-cognitive training on the functional and cognitive capacity of older people with mild cognitive impairment: a randomized controlled trial. BMC Med. 2024 Jul 8;22(1):281. doi: 10.1186/s12916-024-03469-x. PMID 38972988